CLINICAL TRIAL: NCT00468338
Title: Correlation Between the Severity of Mental Retardation and BIS in Mentally Retarded Patients Undergoing Dental Rehabilitation
Brief Title: Correlation BIS Scores Mentally Retarded Patients
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: 0120060266
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2015-04

CONDITIONS: Mental Retardation
Keywords: general anesthesia; dental rehabilitation; mental retardation
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BIS monitor used for all subjects: BIS monitor applied to all subjects
  Interventions: Device: BIS monitor

INTERVENTIONS:
Device: BIS monitor — BIS monitor measures the depth of anesthesia and was used in the entire group

SUMMARY:
The BIS monitor is a tool which assists anesthesiologists in monitoring the depth of anesthesia or level of anesthesia. The study doctors would like to see if it is useful tool for patients who are mentally challenged and require anesthesia.

DETAILED DESCRIPTION:
General endotracheal tube anesthesia (GETA) is administered for mentally retarded patients that need dental rehabilitation. GETA is done, in all patients, with routine monitoring of electrocardiography, blood pressure recording, pulse oximetry and end-tidal capnography. These measurements are also used indirectly to determine the depth of anesthesia and the anesthetic is titrated to prevent awareness during surgery and any subsequent recall (1). In addition, a recently introduced functional electroencephalography (EEG)-based awareness monitor directly analyzes the brain wave pattern during anesthetic delivery and aids the anesthesiologist in maintaining the ideal depth of anesthesia. The EEG based monitor serves to prevent awareness and recall due to light anesthesia or prolonged recovery following deep anesthesia (2). This instrument, named the Bispectral Index Scale (BIS) monitor, is non-invasive and is approved by the Food & Drug Administration. However, the BIS monitor is not being used routinely during the anesthetic management of mentally retarded patients due to a belief that such monitoring would be inaccurate in this cohort of patients (3). This assumption lacks scientific validation. Our trial will investigate the usefulness of BIS monitoring in mentally retarded patients and document any correlation between the severity of mental retardation and BIS scoring during various phases of anesthesia, such as awake status and sedation prior to anesthesia, induction and maintenance of anesthesia, and emergence and recovery from anesthesia. The anesthetic protocol will be standardized and the anesthetic management will not deviate from routine practice. The adjuvant therapies for infection prophylaxis and pain control will be administered in the usual fashion.

ELIGIBILITY:
Inclusion Criteria:

* mentally retarded persons ages 12 to 65 undergoing dental rehabilitation

Exclusion Criteria:

* patients who are pregnant parents/and or legal guardians who do not wish to give consent

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: mentally retarded persons ages 12 to 65 ubdergoing dental rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2006-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rex Ponnudurai, MD, Principal Investigator — University of Medicine and Dentistry of New Jersey
Locations (1):
- UMDNJ University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dahaba AA. Different conditions that could result in the bispectral index indicating an incorrect hypnotic state. Anesth Analg. 2005 Sep;101(3):765-773. doi: 10.1213/01.ane.0000167269.62966.af. PMID 16115989